CLINICAL TRIAL: NCT03286361
Title: Belgo-France Physician-initiated Trial Investigating the BeGraft Peripheral Plus Stent Graft System for the Treatment of Iliac Lesions (TASC A, B, C and D)
Brief Title: Clinical Trial Investigating the BeGraft Peripheral Plus Stent Graft System for Iliac Lesion Treatment
Acronym: BeGraft+PMCF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ID3 Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID3-20170711
Record Dates: First submitted 2017-09-15; First posted 2017-09-18 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BeGraft Peripheral + Stent Graft System (Experimental): Patients treated with the BeGraft Peripheral Plus Stent Graft System
  Interventions: Device: BeGraft Peripheral Plus Stent Graft System

INTERVENTIONS:
Device: BeGraft Peripheral Plus Stent Graft System — Patients will be treated with the BeGraft Peripheral Plus Stent Graft System

SUMMARY:
The BeGraft Plus PMCF Trial investigates the efficacy of the BeGraft Peripheral Plus Stent Graft System in the treatment of iliac stenotic or occlusive lesions (TASC A, B, C and D). An expected total of 20 patients with TASC A and B lesions and an expected total of 50 patients with TASC C and D lesions will be treated. The lesion is located within the native Iliac arteries. Prior to stenting with the BeGraft Peripheral Plus Stent Graft System, pre-dilatation can be performed according to the physician's discretion. Also post-dilatation can be performed according to the physician's discretion. Patients will be invited for a follow-up visit at 1, 6, 12, 24 and 36- month post-procedure. The primary efficacy endpoint of the study is the primary patency at 12 months. The primary safety endpoint is the freedom of periprocedural Serious Adverse Events (SAEs). Secondary endpoint include primary patency rate at 1, 6, 24, and 36-month, stent graft occlusion rate at pre-discharge,1, 6, 24, and 36 month follow-up, anke-brachial index (ABI) at 1, 6, 12, 24 and 36-month follow-up, amputation rate at 1, 6, 12, 24 and 36-month follow-up, performance success rate, freedom from target lesion revascularization (TLR), technical success and clinical success at 1, 6, 12, 24 and 36-month follow-up. The extension in the Begraft Plus protocol is being made to evaluate the long-term safety and efficacy of the BeGraft Peripheral Plus Stent Graft.

DETAILED DESCRIPTION:
The objective of this clinical investigation is to evaluate, in a controlled setting, the long-term safety and efficacy of the BeGraft Peripheral Plus Stent Graft System in clinical settings post CE-certification when used according to the indications of the IFU with focus on the treatment of complex TASC A, B, C and D iliac lesions.

Patients will be selected based on the investigator's assessment, evaluation of the underlying disease and the eligibility criteria. The patient's medical condition should be stable, with no underlying medical condition which would prevent them from performing the required testing or from completing the study. Patients should also be geographically stable, willing and able to cooperate in this clinical study and remain available for long-term follow-up. A patient is considered enrolled in the study after obtaining the patients informed consent, if there is full compliance with the study eligibility criteria and after successful guidewire passage through the study target lesion.

Prior to the index procedure the following tests and clinical data will be collected: informed consent for data collection, demographics, medical history, medication record, physical examination, clinical category of chronic limb ischemia (Rutherford category) and resting ankle-brachial index (ABI).

During the procedure, the vascular access can be achieved to the investigator's standard clinical practice. After successful lesion passage, diagnostic angiography of the lesion area and distal run-off is performed and angiographic measurements (vessel diameter, percentage stenosis and lesion length) are collected. At the physician's discretion, the patient receives at least 1 BeGraft Peripheral Plus Stent Graft System. Pre- and post-dilatation are according to the physician's discretion. No other adjunctive therapies (atherectomy, laser) are allowed. The complete iliac vasculature should be treated in one single session, staged interventions are not allowed. All outflow-limiting lesions must be treated according to the hospital treatment standard.

The regular follow-ups are necessary to monitor the condition of the patient and the stent/procedure. Patients will be invited for a follow-up visit at 1, 6, 12, 24 and 36 months after the index procedure. The following data will be collected during these follow-up visit: medication record, physical examination, rutherford categorization, ABI and color flow doppler ultrasound.

ELIGIBILITY:
General inclusion criteria

* Corresponding to the Conformité Européenne (CE)-mark indications/contra-indications and according to the current medical guidelines for minimally invasive peripheral interventions.
* Patient presenting with a stenotic or occlusive lesion at the iliac arteries suitable for stenting (on indication for primary stenting, based on the discretion of the investigator)
* Patient presenting a score from 2 to 5 following Rutherford classification
* Patient is willing to comply with specified follow-up evaluations at the specified times for the duration of the study
* Patient is >18 years old
* Patient (or their legal representative) understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* Patient is eligible for treatment with the BeGraft Peripheral Plus Stent Graft System (Bentley)
* Patient is treated as emergency case (ruptures, perforations, aneurysms and fistulae)

Angiographic inclusion criteria:

* The target lesion has angiographic evidence of stenosis or restenosis > 50% or occlusion which can be passed with standard guidewire manipulation
* There is angiographic evidence of a patent Common and Deep Femoral Artery
* The target lesion is either a modified TASC-II class A, B, C or D lesion with one of the listed specifications:

  o Type A lesions
* Unilateral or bilateral stenosis of the Common Iliac Artery
* Unilateral or bilateral single short (≤3 cm) stenosis of the External Iliac Artery

  o Type B lesions
* Unilateral Common Iliac Artery occlusion
* Single or multiple stenosis totaling 3-10 cm involving the External Iliac Artery not extending into the Common Femoral Artery
* Unilateral External Iliac Artery occlusion not involving the origins of Internal Iliac Artery or Common Iliac Artery

  o Type C lesions
* Bilateral Common Iliac Artery occlusions
* Bilateral External Iliac Artery stenoses 3-10 cm long not extending into the Common Femoral Artery

  o Type D lesions
* Unilateral occlusions of both Common Iliac and External Iliac Artery
* Diffuse disease involving the aorta bifurcation
* Bilateral occlusions of External Iliac Artery

Exclusion Criteria:

* PTA is technically not possible (not feasible to access the lesion or a defect with the guidewire or balloon catheter)
* Presence of an aneurysm immediately adjacent to the site of stent implantation
* Stenosis distal to the site of stent implantation
* Lesions in or adjacent to essential collaterals(s)
* Lesions in locations subject to external compression
* Heavily calcified lesions resistant to percutaneous transluminal angioplasty (PTA)
* Patients with diffuse distal disease resulting in poor stent outflow
* Patients with a history of coagulation disorders
* Patients with aspirin allergy or bleeding complications and patients unable or unwilling to tolerate anticoagulant/antiplatelet therapy and/or non-responders to anticoagulant/antiplatelet therapy
* Fresh thrombus formation
* Patients with known hypersensitivity to the stent material (L605) and or polytetrafluoroethylene (PTFE)
* Previously implanted stent(s) at the same lesion site
* Reference segment diameter is not suitable for the available stent design
* Untreatable lesion located at the distal outflow arteries
* Use of alternative therapy (e.g. atherectomy, cutting balloon, drug-coated balloon (DCB), laser, radiation therapy) as part of the index procedure
* Patients refusing treatment
* Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated
* Patients who exhibit persistent acute intraluminal thrombus of the proposed lesion site
* Patients with a history of prior life-threatening contrast medium reaction
* Patients with uncorrected bleeding disorders
* Female patient with child bearing potential not taking adequate contraceptives or currently breastfeeding
* Life expectancy of less than twelve months
* Any planned surgical intervention/procedure within 30 days of the study procedure
* Any patient considered to be hemodynamically unstable at onset of procedure
* Patient is currently participating in another investigational drug or device study that has not completed the entire follow up period.
* The target lesion is either a modified TASC-II class B, C or D lesion with aortic or common femoral lesion involvement:

  o Type B lesions
* Short (≤3 cm) stenosis of infrarenal aorta

  o Type C lesions
* Unilateral External Iliac Artery stenosis extending into the Common Femoral Artery
* Unilateral External Iliac Artery occlusion that involves the origins of the Internal Iliac and/or Common Femoral Artery
* Heavily calcified unilateral External Iliac Artery occlusion with or without involvement of origins of the Internal Iliac and/or Common Femoral Artery

  o Type D lesions
* Infra-renal aortoiliac occlusion
* Iliac stenoses in patients with an Abdominal Aortic Aneurysm (AAA) requiring treatment and not amenable to endograft placement or other lesions requiring open aortic or iliac surgery
* Diffuse multiple stenoses involving the unilateral Common Iliac, External Iliac and Common Femoral Artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-11-29 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Primary patency at 12 months | 12 months
  Freedom from >50% restenosis as indicated by an independently verified duplex ultrasound peak systolic velocity ratio (PSVR) <2.5 in the target vessel with no target lesion revascularization within 12 months.
Periprocedural Serious Adverse Events (SAEs) | 30-days post-procedure
  Periprocedural SAEs up to 30-days post-procedure, as defined according to the International Organization of Standardization (ISO) guidelines: ISO 14155:2011

SECONDARY OUTCOMES:
Primary patency rate | 1-, 6-, 24- and 36-months post-procedure
  Freedom from >50% restenosis as indicated by an independently verified duplex ultrasound peak systolic velocity ratio (PSVR) <2.5 in the target vessel with no target lesion revascularization within 12 months.
Stent graft occlusion rate | Pre-discharge, 1-, 6- 12-, 24-, and 36-month follow-up
  Occlusion of the stent graft system
Ankle-brachial index (ABI) | 1-, 6-, 12-, 24-, and 36-month follow-up
  ABI at follow-up compared with the baseline ABI
Amputation rate | 1-, 6-, 12-, 24-, and 36-month follow-up
  Any amputation above the knee
Performance success rate | Baseline
  Successful in sealing acute perforation or rupture, in treating aneurysms and fistulae of restoration of blood flow
Freedom from target lesion revascularization (TLR) | 1-, 6-, 12-, 24-, and 36-month follow-up
  Freedom from a repeated intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5mm proximal and distal to the treated lesion edge
Technical success | Index procedure
  Ability to achieve final residual angiographic stenosis no greater than 30%
Clinical success | 1-, 6-, 12-, 24-, and 36-month follow-up
  Improvement of Rutherford classification compared to the pre-procedure Rutherford classification

CONTACTS AND LOCATIONS:
Overall Officials: Koen Deloose, MD, Study Director — ID3 Medical
Locations (9):
- Belgium (8):
  - O.L.V. Hospital, Aalst
  - ZNA, Antwerp
  - Imelda Hospital, Bonheiden
  - A.Z. Sint-Blasius, Dendermonde
  - ZOL, Genk
  - az Groeninge, Kortrijk
  - RZ Heilig Hart, Tienen
  - AZ Jan Portaels, Vilvoorde
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No